CLINICAL TRIAL: NCT00313794
Title: Phase 2, Single Arm Study Of Ticilimumab In Patients With Refractory Metastatic Adenocarcinoma Of The Colon Or Rectum
Brief Title: Study of Ticilimumab in Patients With Metastatic Colorectal Cancer Whose Disease Had Progressed After Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3671014
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): single arm
  Interventions: Drug: CP-675,206

INTERVENTIONS:
Drug: CP-675,206 — 15 mg/kg IV q 3 months for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Other Names: ticilimumab, tremelimumab

SUMMARY:
This study is for patients with metastatic adenocarcinoma arising from the colon or rectum who have received treatment(s) for metastatic disease with subsequent disease progression. Patients who are intolerant to treatment(s) are also included. This is a study for good performance status colorectal cancer patients who have exhausted standard therapy options.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of metastatic, progressive disease following standard therapies.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

Exclusion Criteria:

* Known brain metastases or uncontrolled pleural effusions.
* History of chronic inflammatory or autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To assess the best overall response rate per RECIST (BRR) in patients with metastatic adenocarcinoma of the colon or rectum treated with CP-675,206 . | 18 months

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of CP-675,206 in this population. | 18 mos
To identify any human anti human antibody (HAHA) response to CP-675,206 . | 3 yrs
To identify potential relationships between polymorphisms in the Cytotoxic T lymphocyte-associated antigen 4 (CTLA4), Fcgamma receptor IIa (FcgRIIa), IgG2a genes with safety and/or immune response of patients treated with CP-675,206. | 3 yrs
To assess additional evidence of anti-tumor activity as measured by duration of response, progression-free survival and overall survival. | 2 yrs
To obtain pharmacokinetic (PK) data to be evaluated in a future meta analysis of CP-675,206 pharmacokinetics. | 3 yrs

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Research Site, Bessemer, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, San Francisco, California
  - Research Site, New York, New York
- Canada (2):
  - Research Site, Lévis, Quebec
  - Research Site, Québec, Quebec